CLINICAL TRIAL: NCT03480672
Title: Postoperative Adjuvant Radiochemotherapy (aRCH) With Cisplatin (C) Versus aRCH With C and Pembrolizumab (P) in Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC); Multicenter Randomized Phase II Study Within the German Interdisciplinary Study Group of German Cancer Society (IAG KHT); Pembro-Adjuvant-highRisk
Brief Title: Postoperative aRCH With Cisplatin Versus aRCH With Cisplatin and Pembrolizumab in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Andreas Dietz, Prof. Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADRISK
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Chemoradiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab + aRCH (Experimental): Application of pembrolizumab, i.v., in 3-week cycle (q3w) 200 mg, in combination with standard treatment (adjuvant radio-chemotherapy aRCH)
  Interventions: Drug: Pembrolizumab 25 MG/1 ML Intravenous Solution [KEYTRUDA]; Other: adjuvant radiochemotherapy
- aRCH (Active Comparator): adjuvant radio-chemotherapy (aRCH)
  Interventions: Other: adjuvant radiochemotherapy

INTERVENTIONS:
Drug: Pembrolizumab 25 MG/1 ML Intravenous Solution [KEYTRUDA] — intravenous application, 12 months, in 3-week cycle (q3w) 200 mg
  Arms: Pembrolizumab + aRCH
Other: adjuvant radiochemotherapy — adjuvant radiochemotherapy with cisplatin

SUMMARY:
This trial evaluates the addition of pembrolizumab to standard postoperative adjuvant radiochemotherapy in the treatment of patients with locally advanced intermediate and high risk head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

1. Macroscopically complete resection of newly diagnosed (not recurrent, not secondary primary) advanced squamous-cell carcinoma arising in the oral cavity, oropharynx, larynx, or hypopharynx
2. Advanced stage III, IVA/B HNSCC according to the TNM classification version 7th edition (Note! The 8th edition will not be used, please adhere to the national cancer institute guidelines)
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; performance status allows adjuvant chemo radiation with cisplatin.
4. Had either intermediate or high-risk characteristics, i.e. any or all of the following:

   * histologic evidence of invasion of two or more regional lymph nodes
   * extracapsular extension of nodal disease,
   * microscopically involved mucosal margins of resection (R1) or margins of resection < 5mm (R0)
5. Had pathological histologic assessment of p16 (only oropharyngeal carcinoma)
6. Be > 18 years of age
7. Written informed consent
8. Demonstrate adequate organ function
9. Female subject of childbearing potential should have a negative pregnancy test within 3 days prior to receiving the first dose of study medication.
10. Female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication.
11. Reproductive male subjects must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

1. Concurrent participation in any other interventional clinical trial or participation in any other interventional trial within one month before enrolment into this trial.
2. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before enrolment into this trial.
3. Known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to Pembrolizumab or comparable medicinal products or any of its excipients.
5. Prior anti-cancer monoclonal antibody (mAb) therapy within one month before enrolment into this trial or who has not recovered (i.e., ≤ Grade 1 (NCI CTCAE Grade) at baseline) from adverse events due to agents administered more than one month earlier.
6. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within one month before enrolment into this trial or who has not recovered (i.e., ≤ grade 1 (NCI CTCAE Grade) at baseline) from adverse events due to a previously administered agent.

   1. Note: Subjects with ≤ Grade 2 (NCI CTCAE Grade) neuropathy are an exception to this criterion and may qualify for the study.
   2. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Active autoimmune disease that has required systemic treatment in the past 2 years prior to enrolment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Evidence of interstitial lung disease or history of (non-infectious) pneumonitis that required steroids within the last 6 months before enrolment into this trial, or current pneumonitis.
10. Active infection requiring systemic therapy.
11. Suspected lack of compliance
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the baseline visit through 120 days after the last dose of trial treatment.
13. HIV, HBV or HCV infection
14. Application of a live vaccine within one month of enrolment.
15. Hypersensitivity to cisplatin or any of its excipients
16. Any potential relationship to the investigator/his deputy or to medical staff of the study team, to the coordinating investigator or is an employee of the study sit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | 24 months
  time from randomization to the first event (i.e. locoregional or distant recurrence, initiation of a new anti-cancer treatment death from any cause)

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Dietz, Prof. Dr., Principal Investigator — University Leipzig
Locations (16):
- Germany (16):
  - Charité - Universitätsmedizin Berlin; Klinik für Radioonkologie und Strahlentherapie CVK, Berlin
  - Charité - Universitätsmedizin, CVK und CCM, Klinik für Hals-Nasen-Ohrenheilkunde, Berlin
  - Klinikum Bielefeld, Onkologie/Hämatologie/ Palliativmedizin, Bielefeld
  - Universitätsklinikum Bonn; Med. Klinik III / ZIM, Hämatologie/Onkologie, Bonn
  - Universitätsklinikum Düsseldorf, Klinik für Strahlentherapie und Radiologische Onkologie, Düsseldorf
  - Helios Klinikum Erfurt GmbH, Klinik für Hals-Nasen-Ohrenheilkunde, Erfurt
  - Universitätsklinikum Essen, Klinik und Poliklinik für Strahlentherapie, Essen
  - Kath. Marienkrankenhaus gGmbH, Zentrum für Innere Medizin Hämatologie/Onkologie, Hamburg
  - Universitätsklinikum Jena, Klinik für Hals-Nasen-Ohrenheilkunde, Jena
  - Department of Head Medicine and Oral Health, University of Leipzig, Leipzig
  - UNIVERSITÄTSKLINIKUM Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Mannheim, Hals-Nasen-Ohren Klinik, Mannheim
  - Ernst von Bergmann Klinikum Potsdam, Zentrum für Hämatologie, Onkologie und Strahlenheilkunde, Klinik für Hämatologie und, Potsdam
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Strahlentherapie, Regensburg
  - Klinikum Stuttgart - Katharinenhospital, Klinik für Radioonkologie und Strahlentherapie, Stuttgart
  - Universitätsklinikum Würzburg; Klinik und Poliklinik für Strahlentherapie, Würzburg

IPD SHARING:
Plan to Share IPD: No